CLINICAL TRIAL: NCT00784004
Title: Investigation of Efficiency of Breathing With Different Breathing Patterns in Healthy Volunteers and Patients With Respiratory Failure
Brief Title: Investigation of Efficiency of Breathing With Different Breathing Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Assistant Professor of Anesthesia, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-P-001371
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Physiology; Respiratory Insufficiency; Breathing Patterns
Keywords: breathing patterns,; unidirectional breathing,; mask ventilation,; respiratory physiology
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volunteers (Other): Ten healthy volunteers
  Interventions: Other: Breathing Patterns
- Patients (Other): Sixteen patients with respiratory insufficiency
  Interventions: Other: Breathing Patterns

INTERVENTIONS:
Other: Breathing Patterns — All subjects will breathe in four different breathing patterns which are provided by specific masks. Patterns are as the following:
  1. Breathing in through the nose only and out through the mouth only
  2. Breathing in through the mouth only and out through the nose only
  3. Breathing in and out through the nose only
  4. Breathing in and out through the mouth only

SUMMARY:
Our aim in this study is to investigate the efficiency of the breathing with different breathing patterns. Ten volunteers and twenty patients having respiratory problems will be coached on their breathing through specific masks which will provide four different breathing patterns. These patterns will be 1) Breathing in through the nose only and out through the mouth only 2) Breathing in through the mouth only and out through the nose only 3) Breathing in and out through the nose only 4) Breathing in and out through the mouth only The data obtained from volunteers and patients will be compared within and between the groups.

ELIGIBILITY:
Inclusion Criteria:

* For healthy subjects:

  1. Ten healthy adult (> 18 years of age) volunteers will be recruited from the MGH main campus through intra-hospital e-mail broadcasting. Subjects with the following issues will be excluded from the study.
* For patients with respiratory insufficiency:

  1. Twenty adult (> 18 years of age) patients will be recruited. These patients will be either patients in acute respiratory failure resulting from COPD exacerbation breathing spontaneously only receiving nasal oxygen admitted to the medical floors of the MGH; or patients with diagnosed stable COPD on home oxygen therapy seen by pulmonary physicians in the outpatient clinics or coming to the MGH as study subjects.

Exclusion Criteria:

* For healthy volunteers:

  1. Subjects with facial deformity, heavy beard or moustache which prevents good seal between the mask and the face;
  2. Subjects who have claustrophobia and cannot wear the mask.
* For patients with respiratory insufficiency:

  1. Patients with facial deformity, heavy beard or moustache which prevents a good seal between the mask and the face;
  2. Patients who have claustrophobia and cannot wear the mask.
  3. Patients who are hemodynamically unstable.
  4. Patients requiring continuous noninvasive positive pressure ventilation or endotracheal intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determining the anatomic dead space change at variable tidal volumes with four different breathing patterns (nose-in and nose-out, mouth-in and mouth-out, nose-in and mouth-out, mouth-in and nose-out) in healthy volunteers. | 3 months
Comparing the efficiency of CO2 removal at given minute ventilations with the four different breathing patterns in patients with chronic respiratory failure. | 6 months

SECONDARY OUTCOMES:
Comparing the efficiency of the study mask which forces subjects to breathe in a manner similar to pursed lip breathing and a regular facemask in healthy volunteers and patients with respiratory failure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Respiratory Care Laboratory, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sulemanji DS, Bao F, Jiang Y, Kacmarek RM. A unidirectional breathing pattern improves breathing efficiency in subjects with severe COPD. Respir Care. 2014 Oct;59(10):1487-93. doi: 10.4187/respcare.02899. Epub 2014 Apr 29. PMID 24782549